CLINICAL TRIAL: NCT03340714
Title: A Pilot Study Investigating the Feasibility of ADAMM (Automated Device for Asthma Monitoring and Management) in Combination With Electronic Patient-Reported Outcomes in Adult Patients With Lung Cancer
Brief Title: Automated Device for Asthma Monitoring and Management in Monitoring Adults With Lung Cancer Undergoing Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Health Care Originals, Inc. (Unknown)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 17P.209; JT 10294 (Other: JeffTrial Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-01

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Device Feasibility (ADAMM): Patients wear the Automated Device for Asthma Monitoring and Management (ADAMM) from the time of computed tomography (CT) simulation for radiation therapy (RT) planning throughout the entire RT course and for 4 weeks post-RT
  Interventions: Device: Monitoring Device

INTERVENTIONS:
Device: Monitoring Device — Wear ADAMM

SUMMARY:
This pilot early phase I trial studies the Automated Device for Asthma Monitoring and Management in monitoring adult patients with lung cancer who are undergoing radiation therapy. The Automated Device for Asthma Monitoring and Management may provide useful information to doctors to help monitor adult patients with lung cancer and diagnose certain conditions earlier than traditional means.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine compliance with the Automated Device for Asthma Monitoring and Management (ADAMM) device in patients receiving radiation therapy (RT) for lung cancer.

SECONDARY OBJECTIVES:

I. Evaluate feasibility of recruitment, acceptability of the ADAMM device, and compliance with electronic patient-reported outcomes (ePROs) in this patient population

ELIGIBILITY:
Inclusion Criteria:

* Patients are capable of giving informed consent
* Patients are eligible to be treated with RT and plan to start treatment
* Patients have either metastatic or non-metastatic lung cancer as defined in history and physical
* Patients must be able to read or speak English
* Women of reproductive potential should have a negative serum or urine pregnancy test within one week prior to radiation planning CT scan

Exclusion Criteria:

* Patients who cannot read or speak English
* Patients who are not candidates for RT treatment
* Women of childbearing potential who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic and non-metastatic lung cancer being treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Percentage of hours per day that patients wear the Automated Device for Asthma Monitoring and Management device | Up to 4 weeks post-radiation therapy
  The compliance rate along with a one-sided exact 95% confidence interval will be estimated.
Percentage of days per study period that patients wear the Automated Device for Asthma Monitoring and Management device | Up to 4 weeks post-radiation therapy
  The compliance rate along with a one-sided exact 95% confidence interval will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/